CLINICAL TRIAL: NCT01270061
Title: Project Wellness: Increasing HIV Testing Among West African Immigrants
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We did not receive proper funding to complete this study
Sponsor: North Bronx Healthcare Network (Other)
Responsible Party: Principal Investigator, Yvette Calderon,MD, MS, Professor of Clinical Emergency Medicine, North Bronx Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2010-587
Record Dates: First submitted 2011-01-03; First posted 2011-01-05 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes; Hypertension; HIV
Keywords: HIV testing; black Africans; immigrants; health screening
MeSH Terms: conditions — Diabetes Mellitus; Hypertension | interventions — HIV Testing

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIV testing (Active Comparator): Group 1 (Control) is the current standard of care in HIV testing. A trained counselor provides required information to obtain informed consent for HIV testing and provides rapid HIV testing on site.
  Interventions: Behavioral: HIV testing
- General Health Screening (Experimental): In Group 2 (Intervention), a theory-based video is used to obtain informed consent for a free general health screening that includes a blood pressure check, blood glucose measurement, and an HIV test.
  Interventions: Behavioral: General Health Screen

INTERVENTIONS:
Behavioral: HIV testing — HIV education and counseling from a trained Research Assistant and offering of a free rapid, oral HIV test.
  Arms: HIV testing
Behavioral: General Health Screen — A video will provide health education on diabetes, hypertension, and HIV. The video will then offer free blood pressure check, blood glucose measuring, and a free, rapid oral HIV test.
  Arms: General Health Screening

SUMMARY:
Project Wellness is a new intervention that combines the use of culturally-sensitive, video-based education, a general health screening approach, and a community pharmacy setting into one program to improve black African immigrant participation in voluntary HIV testing. The study is divided into three phases: qualitative research; video production; and a feasibility trial. In Phase 1, the investigators will conduct in-depth interviews and focus group discussions with black African participants to obtain insights on overlapping and resonating themes that will help increase participation in HIV testing among black Africans in the Bronx. In Phase 2, data obtained through qualitative work will guide the development of four health education videos. A culturally-tailored educational video on diabetes, hypertension, and HIV will be developed and produced for each gender and in both English and French. In phase 3, the investigators will test the feasibility of a pharmacy-based, culturally-tailored, general health screen that includes rapid HIV testing. The trial will help determine the feasibility of using a computer-based model; recruitment of black Africans in the pharmacies; acceptance of testing; and linking individuals diagnosed with health problems into medical care. A secondary analysis will also determine predictors of refusing to be tested.

DETAILED DESCRIPTION:
Black African immigrants living in the United States have exceptionally high rates of HIV and AIDS. Sub-Saharan Africa remains the epicenter of the global HIV epidemic, accounting for 22.5 of the 33.3 million people living with HIV worldwide. Political, economic, and social instability in many African countries has resulted in an escalating number of Africans migrating to the United States. The number of black African immigrants in the U.S. is growing, having increased 166% between 1990 and 2000. The 1.4 million documented African-born immigrants in the U.S. in 2007 does not account for the many undocumented Africans living in the U.S. Immigrant-related stressors, particularly for undocumented migrants, present challenges to both black Africans and healthcare providers seeking to engage this community in HIV testing and treatment. Characteristically long delays in accessing health services and accepting HIV testing have resulted in a greater proportion of black Africans presenting with an AIDS diagnosis (45%), compared to both U.S.-born non-blacks (25%) and U.S.-born blacks (35%). As the U.S. community of black Africans continues to grow, efforts are needed to reduce the impact of HIV within such marginalized communities.

The lack of culturally sensitive voluntary HIV testing programs has discouraged early diagnoses and treatment for African-born immigrants in the United States. The investigators are developing a new theory-driven HIV testing program that builds on the successful history of developing HIV testing models in the emergency department (ED), but relies on partners from the black African immigrant community to address specific cultural, social, and practical barriers to HIV testing faced by their communities. Traditional methods of HIV testing have not been successful in testing high percentages of black Africans in the U.S. for several reasons including (1) their reluctance to access health care for prevention; (2) their unwillingness to disclose information to their social networks, thus rendering ineffective the CDC-recommended social networking strategies for reaching disaffected populations; (3) the stigma of HIV; and (4) cultural and migrant-specific factors that pose barriers to accessing health care. The investigators propose to partner with black African immigrant community members to identify the cultural and migrant-specific factors that interfere with HIV testing, identify those that characterize the African migrant experience regardless of country of origin, and develop videos that can be used to increase willingness to be tested at community testing sites. The investigators plan to develop and pilot Project Consensus, which will use a trusted community setting - the pharmacy - to establish a permanent site for HIV testing that will engage large numbers of black Africans; increase HIV awareness and eliminate the need to rely on social networks; and reduce stigma by placing HIV testing in the context of a general health screening.

This proposal is based on eight years of research and experience developing and testing BRIEF, a Bronx-based rapid HIV testing program in the ED that utilizes theory-based risk reduction videos and a user-friendly interactive touch screen computer program. The investigators have tested over 53,000 Bronx residents, with high acceptance rates (95%) for adult HIV testing and a high rate (85%) of linking HIV+ patients into specialized medical care. Project Consensus was developed out of recognition that BRIEF does not eliminate important barriers to HIV testing for black African immigrants, a community that suffers disproportionately from the health and social consequences of HIV. Given an increasing emphasis within the U.S. on efficient preventive care, this intervention has the potential to provide an exemplary method for engaging members of immigrant communities in earlier stages of disease.

The study has three phases: Phase 1 consists of interviews and focus groups to obtain community input on social and cultural barriers to testing. This input will frame the content of a health education video, as well as the creation of an effective HIV testing program. Phase 2 will develop the HIV testing intervention. Phase 3 is a feasibility trial to prepare for a future randomized controlled trial. An advisory board composed of a diverse group of African community leaders will inform and guide all three phases. There are three specific aims:

1. Use individual interviews and focus groups to identify specific barriers to HIV testing and assess appropriate methods to increase participation in voluntary HIV testing among black African immigrants;
2. Develop a theory-based HIV video to educate and encourage black African immigrants to get tested;
3. Establish the feasibility of the intervention in a community pharmacy that places HIV testing in a general health context, as determined by: standard deviation for the primary outcome of HIV testing rates, use of a computer-based model; recruitment of black Africans in the pharmacies.

   1. Determine the percentage of individuals diagnosed with one of three chronic illnesses linked to care and determine predictors of those that refuse testing.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older
* African-born

Exclusion Criteria:

* unable to understand the consent process
* known HIV status
* tested within the past 3 months
* language other than English or French

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2015-03 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
HIV testing rate | up to 1 hour
  rate of participation in voluntary rapid oral HIV test in each group

SECONDARY OUTCOMES:
Health Knowledge | up to 1 hour
  Change in knowledge of diabetes, hypertension, and HIV.
Risk perception | up to 1 hour
  Change in participants' score on a validated health risk perception measure
Linkage to care | up to one year
  Proportion of positively-screened participants that attend follow-up specialized medical care.

CONTACTS AND LOCATIONS:
Overall Officials: Yvette Calderon, MD, MS, Principal Investigator — North Bronx Healthcare Network
Locations (1):
- Community Bronx, The Bronx, New York, United States